CLINICAL TRIAL: NCT00743769
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Response Phase 1 Study of the Safety and Tolerability of the Intravenous Administration of Thymosin Beta 4 and Its Pharmacokinetics After Single and Multiple Doses in Healthy Volunteers
Brief Title: A Phase 1 Safety Study of the Intravenous Administration of Thymosin Beta in Healthy Volunteers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study never initiated due to contract manufacturing issues
Sponsor: RegeneRx Biopharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RGN-MI-101
Record Dates: First submitted 2008-08-27; First posted 2008-08-29 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Myocardial Infarction; Myocardial Ischemia
Keywords: Myocardial Infarction; Myocardial Ischemia; Myocardial Diseases; Infarction
MeSH Terms: conditions — Myocardial Infarction; Myocardial Ischemia; Cardiomyopathies; Infarction | interventions — thymosin beta(4)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Active Comparator): Thymosin Beta 4
  A single bolus injections of ascending doses of 42 mg, 140 mg, 420 mg or 1,260 QD (once a day)
  Interventions: Drug: thymosin beta 4
- 1 (Placebo Comparator): Placebo A single bolus injection of 0.0 mg QD of thymosin beta 4
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: thymosin beta 4 — Single bolus injections of ascending doses of 42 mg, 140 mg, 420 mg or 1,260 QD of thymosin beta 4
  Arms: 2
Other: Placebo — Single bolus injections of ascending doses of 0.00 mg QD of thymosin beta 4
  Arms: 1

SUMMARY:
The purpose of this study is to determine whether the intravenous administration of single- and multiple-ascending doses of Thymosin Beta 4 is safe and tolerable in healthy volunteers.

DETAILED DESCRIPTION:
The cardio-protective effect of Tβ4 treatment was shown in a permanently ligated mouse model.The authors demonstrated that systemic Tβ4 treatment (intraperitoneal, intracardiac, or i.p. plus intracardiac) every third day enhanced early myocyte survival and significantly improved cardiac function. Several weeks after the heart attack, it was evident that mice treated with Tβ4 had less muscle damage and stronger hearts compared with mice treated with placebo. Specifically, Tβ4 treatment significantly improved fractional shortening by about 60% and ejection fraction by about 100% and myocardial salvage by about 53% when compared with controls.

ELIGIBILITY:
Inclusion Criteria:

* In good health with no underlying medical condition that, according to the Investigator, would place a subject at risk
* Having given written informed consent

Exclusion Criteria:

* Evidence of any malignancy
* Use of any tobacco product within 7 years of study entry
* Pregnant or lactating women
* History of drug abuse
* Clinically significant abnormal screening ECG
* Abnormal vital signs
* Use of systemic steroidal therapy), immunotherapy, cytotoxic, chemotherapy or any investigational drug or device within 30 days of study entry. Topical steroids are allowed
* Women, 40 years of age and above, who have not had a mammography within one year of study entry
* Men and women, 50 years of age and above, who have not had a sigmoidoscopy within 5 years and colonoscopy within 10 years of study entry

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-04; Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Evaluate safety parameters in single-ascending doses of Tβ4(42 mg, 140 mg, 420 mg or 1,260 mg per dose) administered intravenously to healthy volunteers, such as ECG, vital signs,lab tests, etc. | one day

SECONDARY OUTCOMES:
Evaluate pharmacokinetic parameters in single-ascending doses of Tβ4(42 mg, 140 mg, 420 mg or 1,260 mg per dose) administered intravenously to healthy volunteers | one day

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Ruff, MD, Principal Investigator — Healthcare Discoveries LLC
Locations (1):
- Healthcare Discoveries LLC, San Antonio, Texas, United States